CLINICAL TRIAL: NCT04492969
Title: Prospective Observational Study of Failure Patterns in Non-small Cell Lung Cancer Patients Treated With Immune Checkpoint Inhibitors
Brief Title: Prospective Observation of Failure Patterns in NSCLC Treated With ICIs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Other Study IDs: 2019-CSCOBMS
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: NSCLC Stage IV; NSCLC, Recurrent
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
By prospectively observing the time to the best therapeutic effect of non-small cell lung cancer after ICI treatment, the characteristics of lesion distribution when the best therapeutic effect is reached, and the phenotype of disease progression after ICI treatment response, the investigators intended to explore the failure pattern of NSCLC after the once effective ICI treatment. The investigators also aim to evaluate the feasibility and clinical value of radiotherapy for the treatment of oligo-progressive lesions after ICI.

ELIGIBILITY:
Inclusion Criteria (Part I):

* Age between 18 and 75 years.
* ECOG PS 0-1.
* Pathologically confirmed stage IV NSCLC.
* Negative for driver genes including EGFR, ALK, and ROS-1.
* Patients achieved PR or CR after ICI treatment, as defined by RECIST 1.1.
* Patients with complete radiological information of baseline lesions.
* Life expectancy of more than 3 months.
* Ability to understand and willingness to provide the informed consent.

Exclusion Criteria (Part I):

* Severe autoimmune disease or other contradictions to ICI treatment.
* Mixed small cell with non-small cell lung cancer histology.
* Driver gene positive, including EGFR, ALK, and ROS-1.
* Pregnant or lactating women.
* History of any other malignancy.
* Active infection, congestive heart failure, myocardial infarction within the 6 months prior to enrollment, unstable angina pectoris or cardiac arrhythmia.
* Patients receiving immunosuppressive agents,or other investigational treatment. Long-term corticosteroid users are also excluded.
* Mental disorders, drug abuse, and social condition that may negatively impact compliance in the opinion of the investigator.

Inclusion Criteria (Part II, patients with OPD):

* Patients with oligo-progression disease (1-3 progression lesions in 1-2 organs) when developing acquired resistance to ICI.
* Radiotherapy to at least one of the OPD lesions is indicated in the opinion of the investigator. At least one of the irradiated lesion(s) should be evaluable according to RECIST 1.1.
* ECOG PS 0-2.
* Life expectancy of more than 3 months.
* Complete radiological information of all lesions during the follow-up.
* Patients with a prior history of surgery are eligible if they have recovered adequately from the toxicity and/or complications of surgery.
* Adequate bone marrow function within 1 week prior to the enrollment: hemoglobin ≥80g/L, white blood cell (WBC) count ≥ 4.0 * 10 ^ 9/L or neutrophil count ≥ 1.5 * 10 ^ 9/L, and platelet count ≥ 100 * 10 ^ 9/L;
* Ability to understand and willingness to provide the informed consent.

Exclusion Criteria (Part II):

* Secondary malignancy.
* Histology transformation to non-NSCLC.
* Ineligible for radiotherapy in the opinion of the investigator. Or none of the OPD are evaluable by RECIST 1.1.
* ECOG PS 3 or worse.
* Short life expectancy (less than 3 months).
* Unable to provide complete radiological information of lesions.
* Inadequate bone marrow function.
* Cannot understand or unwilling to provide the informed consent.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: stage IV NSCLC developing acquired resistance under ICI treatment.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Oligo-progression disease rate in NSCLC patients developing acquired resistance to ICI treatment. | at least 2 months after ICI treatment.
  Acquired resistance (AR) was defined as disease progression after partial or complete response (PR or CR) to ICI treatment. (by RECIST standard v1.1)
  When observing disease progression in ICI treatment, the number and distribution of progression lesions were recorded.
  Oligo-progression disease (OPD) was defined as 1-3 progression lesions in 1-2 organs. The OPD rate in all AR cases will be calculated.

SECONDARY OUTCOMES:
Overall objective response rate to radiotherapy. | at least 4 weeks after radiotherapy.
  When radiotherapy to at least one of the OPD lesions is indicated in the opinion of the investigator. Overall objective response rate (ORR) to radiotherapy will be recorded. ORR was defined as the proportion of participants with partial response (PR) or complete response (CR) to treatment as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Objective response rate in non-irradiated lesion | at least 4 weeks after radiotherapy.
  Objective response rate (ORR) in Non-irradiated Lesion was defined as the proportion of patients with at least 30% reduction from baseline in the longest diameter of any of non-irradiated target lesions defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 at any time-point from the date of treatment initiation to the date of last follow-up.
Percentage of Participants With Adverse Events | Two years
  Treatment-related adverse events were assessed and graded according to CTCAE v. 5.0.
Overall Survival since AR development. | Two years
  OS was defined as the time from the date of enrollment until death by any cause. Participants still alive at the time of data analysis were censored at the date of last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengfei Zhu, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China